CLINICAL TRIAL: NCT05394129
Title: A Prospective Comparison of SurePath™ Liquid -Based Cytology and Conventional Smear Cytology in Endoscopic Ultrasound-guided Sampling of Esophageal, Gastric, Duodenal Subepithelial Tumors, Periesophageal and Perigastric Lymph Nodes
Brief Title: Diagnostic Accuracy of SurePath™ in EUS-FNA
Status: Terminated | Type: Observational
Why Stopped: Difficulty in recruiting research subjects
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Jeong Cho, Clinical associate professor, Seoul National University Hospital
Other Study IDs: 1902-076-1011
Record Dates: First submitted 2021-09-13; First posted 2022-05-27 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Submucosal Tumor of Gastrointestinal Tract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SurePath™: The subjects are randomly assigned to SurePath™/Conventional test group at a ratio of 1:1.
  In SurePath™ group, subjects who underwent SurePath™ liquid-phase cytology test with the first sample subjected to the conventional smear test with the second sample.
  Interventions: Diagnostic Test: SurePath™
- Conventional: The subjects are randomly assigned to SurePath™/Conventional test group at a ratio of 1:1.
  In conventional test group, those who subjected to the conventional smear test with the first sample, will undergo the SurePath™ liquid cell test with the second obtained sample.
  Interventions: Diagnostic Test: SurePath™

INTERVENTIONS:
Diagnostic Test: SurePath™ — In the liquid-based cytology, a fine-needle aspirated sample is immediately inserted into a container containing a commercially available preservative solution without a separate slide-smearing procedure and immediately after the fine-needle aspiration.

SUMMARY:
It is a prospective randomized controlled study to evaluate the diagnostic accuracy of SurePath™ liquid-based cytology in endoscopic ultrasound-guided sampling.

DETAILED DESCRIPTION:
The SurePath™ has been approved by the FDA since 1997. Investigators want to compare the diagnostic accuracy of SurePath™ liquid based cytology and conventional smear cytology(CSC) in EUS-FNA sampling of esophageal, gastric, duodenal subepithelial tumors, periesophageal and perigastric lymph nodes.

The investigators randomly assigned (1:1) patients to the SurePath™ group or the CSC group. Aspirates from the first needle pass were processed by one method, aspirates from the second pass by the other method, and specimens from the last pass were processed as core biopsy samples. The primary endpoint was the diagnostic efficacy of each method, with the final diagnosis as the gold standard. The aim of this study is to confirm that the SurePath™ is not inferior than the conventional smear test.

ELIGIBILITY:
Inclusion Criteria:

* Patients who signed the agreement after the explanation
* Patients suspected of esophageal, gastric, duodenal subepithelial tumors, periesophageal and perigastric lymph nodes from radiological(CT, MR, ultrasound) or endoscopic examinations.

Exclusion Criteria:

* Those who did not agree with the study
* Patients younger than 19 years of age
* Serious mental patients
* Patients with severe accompanying diseases (ESRD, advanced COPD, severe heart failure, sever mental illness)
* Pregnant women
* If EUS is difficult due to previous surgery (Billroth II or TG with R-en-Y)
* Patient with blood clotting abnormality
* If there is a risk of tract seeding after examination

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients above 19 years of age who underwent EUS-FNA for suspected esophageal, gastric, duodenal subepithelial tumors, periesophageal and perigastric lymph nodes.
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 6 months after randomization
  Pathologic results of the surgical specimen or core needle biopsy will be checked whether it is malignancy or benign. If benign diagnosis is made by combining the results of SurePathTM and conventional smear test, the follow-up period is 6 months and the results of the 6-month follow-up imaging and additional biopsy are checked. The combined results make a final diagnosis and are compared between two groups.

SECONDARY OUTCOMES:
Cytomorphologic feature | 6 months after randomization
  The investigators will evaluate the cytomorphologic features of each method. The investigators plan to investigate whether there are differences in the level of artifacts, the degree of background cleanliness, and tumor cell characteristics such as cellularity.

CONTACTS AND LOCATIONS:
Overall Officials: Han Myung Lee, M.D., Study Director — Fellowship
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No